CLINICAL TRIAL: NCT04552340
Title: Epidemiologic, Clinical and Molecular Characteristics of Patients With Acute Respiratory Failure Affected by 2019-NCOV: A Retrospective-Prospective Cohort Study.
Brief Title: Epidemiologic, Clinical and Molecular Characteristics of Patients With Acute Respiratory Failure Affected by 2019-NCOV.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 2485
Record Dates: First submitted 2020-09-08; First posted 2020-09-17 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-09

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patient with SAR-CoV-2 infection — Study population The study cohort will be enrolled among patients referred to our the Humanitas Research Hospital, the Hospital Cliniche Gavazzeni (Bergamo) hospitals for SARS-CoV-2 screening who will/will not be hospitalized in wards dedicated to COVID-19 patients or admitted to intensive care unit.

SUMMARY:
The main purpose of this study is to identify possible predictor factor of mortality in patients affected by COVID-19 with respiratory failure needing oxygen therapy or ventilatory support. In addiction the study aims to identify factors related to: predisposition to SARS-CoV2 viral infection, different symptoms, response to therapy, predisposition to complications related to the disease. To this end, the haemodynamic parameters and all imaging reports will be evaluated and clinical and laboratory tests as well as cellular and molecular analyzes will be performed in the analyzed patients. In addition, investigations will be carried out on the profile of the alveolar or nasal microbiota and, if possible, of the metabolic products, and estimates on antibody titers.

DETAILED DESCRIPTION:
The study is a cohort study with retrospective-prospective data collection. All the clinical data collected in the study are usually monitored in the clinical practice and no additional clinical exams will be required for the sole purpose of the study.

Patients will be asked consent for the research use of blood and bronchial lavage/residual samples from nasopharyngeal swabs to perform cellular and molecular analyses aimed at better understanding the disease pathogenesis and the individual differences in susceptibility to the disease. These experiments will have no direct impact on the clinical management of patients. It is impossible to detail now all the experiments that will be performed on stored samples. It is possible to anticipate that samples could be used to analyze the immune response by studying immune cells and soluble mediators of the immune response. Moreover, samples will be used to extract nucleic acids to analyze gene expression profiles and DNA variations possibly related with disease susceptibility. Part of the genetic studies could be conducted in other laboratories abroad (i.e. the Institute of Clinical Molecular Biology of the Christian-Albrechts-University of Kiel and the Institute of Clinical Medicine of the University of Oslo) as part of scientific collaborations. In particular, the investigators plan to study the expression levels of molecules known to mediated viral infection, like the Angiotensin converting enzyme 2 (ACE2) and the Transmembrane protease, serine 2 enzyme (TMPRSS2). Genetic variants in these genes, and more in general in other genes in the genome, could be related to susceptibility to the viral infection and/or to the severity of the clinical course of the disease. Therefore, the investigators plan to compare the frequency of genetic variants potentially related with COVID-19 susceptibility/severity in different subgroups of patients, ranging from individuals positive for the virus but asymptomatic to individuals affected by COVID-19 with ARDS requiring admission to ICU. The extension of the analyses that will be performed can't be anticipated as it depends also on the amount of funding that will be available to the study; potentially the entire genome could be analyzed.

Original sepsis and ARDS biomarkers developed at ICH (e.g. PTX3, sIL-1R2, MSF) will be used to address their prognostic potential in COVID-19 patients. PBMC will be analyzed by FACS to investigate the immunophenotype and correlate it to the clinical outcome. Original markers of leukocyte functional activation developed at ICH will be included in the analysis (e.g. IL-1R8, IL-1R2). The residual BAL and rhinopharyngeal swab will be used for microbiota analysis, metabolomics and cytokine measurement. Plasma and saliva/sputum will be used also to test anti-SARS-Cov-2 antibodies (IgM, IgG and IgA) and for microbiota analysis.

In order to better describe the populations of COVID-19 patients treated at our hospital, it is necessary to collect disease outcome data over a short, medium and long-term follow-up process. The investigators aim to understand how disease and intensive treatments affect the lives of recovering patients. In particular, the investigators want to explore the health-related quality of life, the impact of the disease on a psychological level, the residual cardio-respiratory functional capacity and muscle strength. All the tests chosen are common use tests in the follow-up of critically ill patients in particular with acute respiratory distress syndrome.

The health-related quality of the life will be measured with the validated international questionnaire EQ-5D-5L, in its Italian validated form. The questionnaire is attached, and has been authorized for free non-commercial use by the EuroQuol consortium.

As a screening tool to evaluate the presence of psychological symptoms, such as anxiety and depression, the Hospital Anxiety and Depression Scale (HADS) questionnaire will be administered in its Italian version.

The cardio-respiratory functional capacity will be measured with the Six-Minutes Walk Test, following the international guidelines published by the American Thoracic Society.

The single breath count tets will be performed, as well. It consists in the ability to count from zero to twenty after a single maximum inspiration.

Finally, dynamic tests such as the Timed Up-and-Go (TUG) test and the Short physical performance battery (SPPB) test will be performed to evaluate muscle strength, in particular of the lower limbs, the ability to balance while walking and the general mobility of patients. Both the aforementioned tests re internationally validated and are commonly used in the evaluation of the functional reserve of patients in the geriatric and rehabilitation setting. All this tests can be administered to patients during their hospital stay or after their discharge at scheduled appointments.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who underwent to a swab or BAL test for the presence of SAR-CoV-2 infection, aged ≥ 18 years;
* Patients with Acute Respiratory Failure who require ventilatory support / patients admitted to the ICU;
* Patients affected by COVID-19
* Patients infected by SARS-CoV-2.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lack of informed consent according to local procedure per critically ill patients.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2020-03-16 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Mortality predictors in patients with Respiratory Failure who require oxygen therapy in the Intensive Care Unit or ventilatory support. | 1 year
Molecular profile of cell populations present in the BAL at early timepoint during SARS-CoV2 infection to predict severity of disease progression. | 1 year

SECONDARY OUTCOMES:
Type of possible complications such as AKI (Acute Kidney Injury) , infection, shock | 1 year
SARS-CoV2 mechanisms of infection in alveolar macrophages | 3 years
SARS-CoV2 genotypes in a cohort of patients representative of the Lombardy population | 3 years
Number of successful respiratory weaning | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Cecconi, Principal Investigator — Humanitas Research Hospital IRCCS, Rozzano-Milan
Locations (1):
- Humanitas Research Hospital, Rozzano, Milan, Italy